CLINICAL TRIAL: NCT00277706
Title: Impact of Parathyroid Hormone (1-34) on Osseous Regeneration in the Oral Cavity
Brief Title: Impact of Parathyroid Hormone (PTH) on Osseous Cavity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-03
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2009-10-07 (Estimated); Status verified 2009-10

CONDITIONS: Bone Loss; Periodontitis
Keywords: periodontitis; bone regeneration; Parathyroid Hormone; moderate to advanced periodontitis
MeSH Terms: conditions — Bone Diseases, Metabolic; Periodontitis | interventions — Teriparatide; Vitamin D; Calcium

ARMS (2):
- FORTEO (Experimental)
  Interventions: Procedure: Periodontal surgery; Drug: FORTEO; Dietary Supplement: Vitamin D and Calcium
- Placebo (Placebo Comparator)
  Interventions: Procedure: Periodontal surgery; Drug: Placebo; Dietary Supplement: Vitamin D and Calcium

INTERVENTIONS:
Procedure: Periodontal surgery
Drug: FORTEO — parathyroid hormone; self-administration for 6 weeks
  Arms: FORTEO
Drug: Placebo — placebo; self administration for 6 weeks
  Arms: Placebo
Dietary Supplement: Vitamin D and Calcium — PO, QD, for six weeks

SUMMARY:
Parathyroid hormone (PTH) has potent bone-building actions and has been approved for the treatment of osteoporosis as FORTEO by Eli Lilly & Co. Numerous studies have verified its effectiveness in increasing bone mass and potential for PTH to positively impact oral bone. The hypothesis of this study is that patients administered FORTEO along with periodontal (gum) surgery will respond more favorably than patients who receive placebo.

There will be 40 subjects enrolled in this study. All subjects will receive surgical treatment. 20 subjects will receive FORTEO and 20 will receive placebo. Subjects will be assigned to study group randomly. Neither the subjects nor the clinicians will know whether the subject is receiving FORTEO or placebo.

Patients will undergo routine periodontal treatment procedures including periodontal surgery. Starting from 3 days prior to surgery, all subjects will self-administer FORTEO or placebo for 6 weeks. Subjects will be trained for self-administration, a procedure similar to diabetic injections. Patients will also take Vitamin D and Calcium by mouth during this time. Study outcomes will be measured by blood collection; oral fluid sampling; oral x-ray and spine and hip bone density scan; routine periodontal examinations; and an oral health quality of life questionnaire.

Patients of both genders and all ethnicities from age 30-75 years will be included in the study. All ethnicities are eligible for entry into study. No vulnerable populations will be included. Pregnant/breast-feeding women and women of childbearing potential on no contraception will be excluded from the study. Research records will not be linkable to the research subjects. Subjects will be randomly assigned to treatment arms and identified by initials and numbers. Informed consent forms will be used to obtain consent for participation in the study from all subjects prior to enrollment. The Principal Investigator or Co-Investigator will explain the details of study involvement and give subjects ample opportunity to ask questions.

It is anticipated that patients on FORTEO will have greater regeneration with periodontal therapy as compared to control patients.

DETAILED DESCRIPTION:
Parathyroid hormone is an endogenous hormone with potent anabolic and catabolic actions in bone. It has recently been approved for the treatment of osteoporosis and is marketed as FORTEO by Eli Lilly and Company. Numerous studies in humans have validated its use to increase bone mineral density and prevent fractures. Interest has also surfaced in its potential application in the treatment of non-osteoporotic fractures and several animal studies have supported this local application. Little is known regarding its use in treating conditions of the oral cavity, but animal studies suggest that bones of the oral cavity are responsive to the anabolic actions of PTH. Furthermore, a recent study indicated that in a canine model, PTH was effective at reversing periodontal bone loss. Studies from our laboratory indicate that patients with hyperparathyroidism (HPT) do not have an increase in periodontal disease as measured by attachment levels. In fact, in our patient population there was an increase in osseous activity in patients with HPT in the form of tori and exostoses (bony protuberances in the oral cavity). This suggests that increased circulating levels of PTH do not adversely impact the oral cavity. Furthermore, in a wound healing animal model of bone regeneration, we found that regenerating intramembranous bone was more responsive to anabolic actions of PTH than endogenous bone of the vertebrae. These studies highlight the potential for PTH to positively impact osseous healing in the oral cavity in response to periodontal therapy.

The study will be double blinded, and patients will be randomized into one of two treatment groups (FORTEO or placebo once/daily). Patients will self-administer drug on a QD schedule, and take Vitamin D and Calcium, PO, QD, for six weeks. Drug administration will begin three days prior to periodontal surgery. Subjects will be followed at post-op, week 3, week 6, month 3, month 6, month 9, and month 12 visits. Clinical effects will be measured by serum collection, gingival crevicular fluid (GCF) sampling, standard dental radiographs, oral exam including perio probing, oral health quality of life questionnaire, and DEXA scans.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 30 to 75 years
* Sex: Male and female
* Female patients must be postmenopausal (for at least 2 years), surgically sterilized or utilizing one of the following methods of birth control throughout the trial - IUD, diaphragm, Depo-Provera, Norplant, oral contraceptive with condom or spermicidal gel/foam with a condom, or abstinence
* Patients must be able and willing to follow study procedures and instructions
* Patients must have read, understood and signed an informed consent form
* Patients must have localized or generalized, advanced periodontal disease (American Dental Association Class 4)
* Patients must present with at least 10 teeth in the functional dentition
* Each patient must have at least one tooth with the following criteria to enter the study:

  * Periodontal probing depths of > 6 mm to < 14 mm
  * Attachment loss of > 6 mm to < 14 mm
  * Bleeding on probing

Exclusion Criteria:

* Patients under 30 years of age
* Female patients who are pregnant (as determined by positive urine pregnancy test at screening) or lactating, or female patients who are of childbearing potential who are not using hormonal, barrier methods of birth control or abstinence.
* Patients who are using hormonal contraceptives must have started the method not fewer than 30 days prior to the screening examination.
* Patients with metabolic bone diseases such as Paget's disease, hypercalcemia, vitamin D3 abnormalities or any other metabolic bone disease including osteoporosis. (If Vitamin D levels are low (> 20 ng/ml - 24 ng/ml), dietary supplementation will be initiated and levels re-evaluated after 4 weeks and reconsidered for inclusion at that time.)
* Patients with prior radiation treatment, bone metastasis or other skeletal malignancy
* Patients on medications that would affect bone metabolism
* Patients with growth hormone deficiency
* Patients with uncontrolled diabetes, sprue, inflammatory bowel disease or other disorders that would affect calcium absorption.
* Patients who are heavy smokers (> 1 pack/day); Patients on bisphosphonates, including Fosamax
* Patients with any form of kidney disease including kidney stones (urolithiasis and nephrolithiasis); and
* Patients on digitalis therapy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this pilot study is to determine the effect of Forteo (PTH) on periodontal regeneration.

SECONDARY OUTCOMES:
The secondary objectives are to determine the effect of PTH on parameters associated with periodontal health such as attachment level, radiographic bone density and bone height, and gingival crevicular fluid levels of bone active cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie K McCauley, DDS, PhD, Principal Investigator — Professor and Chair
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Bashutski JD, Eber RM, Kinney JS, Benavides E, Maitra S, Braun TM, Giannobile WV, McCauley LK. The impact of vitamin D status on periodontal surgery outcomes. J Dent Res. 2011 Aug;90(8):1007-12. doi: 10.1177/0022034511407771. Epub 2011 May 9. PMID 21555774
- [Derived] Bashutski JD, Eber RM, Kinney JS, Benavides E, Maitra S, Braun TM, Giannobile WV, McCauley LK. Teriparatide and osseous regeneration in the oral cavity. N Engl J Med. 2010 Dec 16;363(25):2396-405. doi: 10.1056/NEJMoa1005361. Epub 2010 Oct 16. PMID 20950166